CLINICAL TRIAL: NCT00961389
Title: Validating a Delirium Prediction Model for Critically Ill Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: M. van den Boogaard, MSc, RN, CCRN, Radboud University Nijmegen Medical Centre
Other Study IDs: 2007/283-2
Record Dates: First submitted 2009-08-17; First posted 2009-08-19 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-08

CONDITIONS: Delirium
Keywords: delirium; critical care; risk factors; prediction; inflammation
MeSH Terms: conditions — Delirium; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- delirious patients: minimal any positive CAM-ICU score during ICU admission
- non-delirious patients: without any positive CAM-ICU score during ICU admission

SUMMARY:
The objective of this study is to determine the incidence of delirium in adults patients who are admitted at the critical care unit of a Dutch University Hospital with the mapping of relevant delirium risk factors The primary aim is to validate the investigators' developed delirium prediction model for critical care patients.

A secondary aim is to find differences between delirious patients and non-delirious patients on different aspects of diagnostics, treatment and care, outcome, length of stay, and inflammation.

According to Dutch law, the need to obtain informed consent was waived by the Committee on Research Involving Human Subjects (CMO) of Nijmegen for this observational study (2007/283).

ELIGIBILITY:
Inclusion Criteria:

* all adult patients (18 years and older) admitted at the critical care unit of our hospital

Exclusion Criteria:

* admitted < 12 hours on ICU
* not able to understand Dutch
* patients with serious hearing and visibility disabilities
* mentally retarded patients
* patients suffering from receptive aphasia
* delirious before admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: tertiary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-09 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
delirium | during admission at the critical care

SECONDARY OUTCOMES:
markers of inflammation | within 24 hours of delirium diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Nijmegen Medical Centre, Critical Care, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] van den Boogaard M, Pickkers P, Slooter AJ, Kuiper MA, Spronk PE, van der Voort PH, van der Hoeven JG, Donders R, van Achterberg T, Schoonhoven L. Development and validation of PRE-DELIRIC (PREdiction of DELIRium in ICu patients) delirium prediction model for intensive care patients: observational multicentre study. BMJ. 2012 Feb 9;344:e420. doi: 10.1136/bmj.e420. PMID 22323509